CLINICAL TRIAL: NCT00245492
Title: Chromocolonoscopy for the Detection of Flat Adenomas in Routine Colorectal Cancer Screening.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: American College of Gastroenterology (Other); Stony Brook University (Other); University of Chicago (Other)
Responsible Party: Charles Kahi, MD, Indiana University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 0508-64; 2005ACG-100CRC
Record Dates: First submitted 2005-10-26; First posted 2005-10-28 (Estimated); Last update posted 2009-01-28 (Estimated); Status verified 2009-01

CONDITIONS: Colon Cancer; Polyp; Adenoma
Keywords: Colonoscopy; Chromoscopy; Prevention
MeSH Terms: conditions — Colonic Neoplasms; Polyps; Adenoma

ARMS (1):
- 1 (Experimental): Chromocolonoscopy
  Interventions: Procedure: Chromocolonoscopy

INTERVENTIONS:
Procedure: Chromocolonoscopy — Indigocarmine dye applied to entire colon to highlight mucosal detail and enhance detection of flat lesions.

SUMMARY:
The proposed research aims to determine the prevalence, size, shape and histology of flat colorectal neoplasms in a cohort of asymptomatic, average-risk individuals presenting for screening colonoscopy. Patients will be randomized to either conventional colonoscopy or chromocolonoscopy, where the entire colon will be sprayed with indigocarmine dye and examined in the usual manner. The primary outcome will be the total number of adenomas detected, with special attention to the subgroup of flat and depressed lesions. To promote the generalizability of the results, neoplasms will be described according to standard Western and Japanese classification schemes.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing screening colonoscopy

Exclusion Criteria:

* Age < 50
* Prior colon resection
* Inflammatory bowel disease
* Prior colonoscopy or sigmoidoscopy
* More than one first-degree relative with colon cancer

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 792 (Estimated)
Dates: Start 2006-05; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Prevalence of adenomas detected by chromocolonoscopy versus standard colonoscopy. | Cross-sectional prevalence of adenomas between the 2 study groups

CONTACTS AND LOCATIONS:
Overall Officials: Charles J Kahi, MD, Principal Investigator — Indiana University School of Medicine, Roudebush VA Medical Center, Indianapolis, Indiana
Locations (3):
- United States (3):
  - Indiana University, Indianapolis, Indiana
  - Roudebush VA Medical Center, Indianapolis, Indiana
  - SUNY Stony Brook, Stony Brook, New York